CLINICAL TRIAL: NCT01657864
Title: WEUSKOP6166: Prevalence of Aseptic Meningitis Among Lamotrigine Users
Brief Title: WEUSKOP6166: Lamotrigine and Aseptic Meningitis
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 117051; WEUSKOP6166 (Other: GSK)
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-07

CONDITIONS: Epilepsy
Keywords: Aseptic Meningitis; Epidemiology; Bipolar Disorder; Lamotrigine; Epilepsy
MeSH Terms: conditions — Epilepsy; Meningitis, Aseptic; Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with aseptic meningitis: All patients of the study population with a record/diagnosis of aseptic meningitis during the study period
  Interventions: Drug: Lamotrigine
- Patients without aseptic meningitis: All patients of the study population without a record/diagnosis of aseptic meningitis during the study period
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine is an anticonvulsant drug used in the treatment of epilepsy and bipolar disorder

SUMMARY:
The objective of the study is to quantify the number of cases of aseptic meningitis among users of Lamotrigine. This study is a cross-sectional study design using data on lamotrigine patients within the Thomson Reuters MarketScan® Commercial database (MarketScan database). The MarketScan database is a US-based insurance claims database representative of a US insured population and includes supplemental datao n Medicare patients. This cross-sectional study will evaluate the number of cases of aseptic meningitis among lamotrigine users during the duration of lamotrigine therapy, with an extended exposure window of 30 days after completing therapy.

The MarketScan® Database is an US insurance claims database that is held in-house at GSK, which can be interrogated to examine rates of prescribing and medical conditions that can be captured via ICD-9 diagnoses codes. The MarketScan database captures person-specific clinical utilization, expenditures, and enrollment across inpatient, outpatient, prescription drug, and carve-out services from a selection of large employers, health plans, and government and public organizations. The annual medical databases include private sector health data from approximately 100 payers. In 2011, there were approximately 35 million patients on the database. The Commercial Claims and Encounters Database represents the medical experience of insured employees and their dependents for active employees, early retirees, COBRA continues, and their dependents insured by employer-sponsored plans (i.e., non-Medicare eligibles). In addition, a linked Medstat Medicare database contains predominantly fee-for-service plan data in insurance plans where both the Medicare-paid amounts and the employer-paid amounts were available and evident on the claims.The data are HIPAA compliant thus all patients have been anonymized.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be using lamotrigine for epilepsy or bipolar disorder.
* Patients must have at least 180 days history on the database prior to the index of lamotrigine use.
* Patients must have medical and pharmacy coverage throughout the study, with no gaps in eligibility.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population for this study includes new user of lamotrigine. To be eligible for this study, Patients were required to use lamotrigine for epilepsy or bipolar disorder. Patients must have at least 180 days history on the database prior to the index of lamotrigine use. Patients must have medical and pharmacy coverage throughout the study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Aseptic meningitis during the period of time the patient is taking lamotrigine | The period at-risk for aseptic meningitis shall begin with the date of the new prescription for lamotrigine and will end 30 days after the last dose of the drug
  The exposure window will be extended by 30 days to be consistent with current pharmacovigilance polices at GSK. Aseptic meningitis coded within this window shall be included in the rate

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline